CLINICAL TRIAL: NCT01652586
Title: Sedation Regimen in Patients Undergoing Cardiac Electrophysiology Study and Ablation : a Comparison Between Dexmedetomidine-remifentanil and Midazolam-remifentanil Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-2011-0008
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Cardiac Arrhythmia
Keywords: cardiac ablation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine-remifentanil (Experimental): intravenous infusion of 0.2-0.7 µg/kg/h of dexmedetomidine after a loading dose of 1 µg/kg over 10 min
  Interventions: Drug: dexmedetomidine-remifentanil
- midazolam-remifentanil (Active Comparator): remifentanil 3.6-7.2 mcg/kg/h midazolam 1-2mg
  Interventions: Drug: midazolam-remifentanil

INTERVENTIONS:
Drug: dexmedetomidine-remifentanil
  Arms: dexmedetomidine-remifentanil
Drug: midazolam-remifentanil
  Arms: midazolam-remifentanil

SUMMARY:
Cardiac ablation is an invasive procedure requiring anesthetic support for immobility and analgesia. Benzodiazepines and opioids are the most commonly used agents, while they are associated with respiratory depression and hypotension. The aim of this study was to compare the effect of remifentanil and dexmedetomidine, which exerts sedative and analgesic effect without serious respiratory depression, with conventional midazolam/remifentanil combination on sedative and analgesic levels in patients undergoing endocardial ablation.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective cardiac ablation for atrial fibrillation

Exclusion Criteria:

* ASA physical status class ≥ 3,
* respiratory disease,
* end stage renal disease,
* illiterate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change of sedation depth | 5 min after study drug adminstration, and every 10 min thereafter
  1. Ramsay sedation score (1 = anxious and agitated, restless; 2 = cooperative, oriented, tranquil; 3 = responsive to verbal commands, drowsy; 4 = asleep, responsive to light stimulation; 5 = asleep, slow response to stimulation; 6 = no response to stimulation)
  2. the bispectral index

CONTACTS AND LOCATIONS:
Overall Officials: Young Lan Kwak, MD, PhD, Principal Investigator — Severance Hospital